CLINICAL TRIAL: NCT04875338
Title: Platelet-rich Plasma, Glucocorticoid, Saline Injection in the Treatment of Lateral Epicondylitis. Randomized Controlled Trial
Brief Title: Injection in the Treatment of Lateral Epicondylitis. Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ahmet Serhat Aydın, asistant doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAD-FR-02
Record Dates: First submitted 2021-04-29; First posted 2021-05-06 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Epicondylitis, Lateral
MeSH Terms: conditions — Tennis Elbow | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: propective randomize
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- saline injection (Active Comparator): 2ml %0.9 NACI(Saline )injection to effected lateral epicondyle
  Interventions: Drug: plate-rich plasma
- platet riched plasma injection (Active Comparator): 2 ml prp )injection to effected lateral epicondyle
  Interventions: Drug: saline (0.9 NACI)
- betametazon injection (Active Comparator): 2 ml betametazon )injection to effected lateral epicondyle
  Interventions: Drug: betametazon

INTERVENTIONS:
Drug: plate-rich plasma — 1ml prp (plate-rich plasma to be prepared with the blood taken from the patient on the day of injection), , while the patient is in the supine position, the affected elbow is 90 flexion and neutral rotation, The non-dominant thumb will be placed at the sensitive point in the lateral epicondyle. The injection will be applied to the point with a 23 g needle. After the injection, the subjects will be taught a stretching exercise of the joint extensors of the wrist and fingers. Subjects will be asked to do this exercise five times in one session, two sessions a day
  Arms: saline injection
Drug: saline (0.9 NACI) — 1 ml saline (0.9 NACI) while the patient is in the supine position, the affected elbow is 90 flexion and neutral rotation, The non-dominant thumb will be placed at the sensitive point in the lateral epicondyle. The injection will be applied to the point with a 23 g needle. After the injection, the subjects will be taught a stretching exercise of the joint extensors of the wrist and fingers. Subjects will be asked to do this exercise five times in one session, two sessions a day
  Arms: platet riched plasma injection
Drug: betametazon — 1 ml betametazon while the patient is in the supine position, the affected elbow is 90 flexion and neutral rotation, The non-dominant thumb will be placed at the sensitive point in the lateral epicondyle. The injection will be applied to the point with a 23 g needle. After the injection, the subjects will be taught a stretching exercise of the joint extensors of the wrist and fingers. Subjects will be asked to do this exercise five times in one session, two sessions a day
  Arms: betametazon injection

SUMMARY:
The aim of the study is to compare the effectiveness of injection techniques in the treatment of elbow lateral epicondylitis. The functional and pain levels of the patients will be evaluated with scores such as DASH, VAS, PRTEE. At the same time, USG imaging will be evaluated before injection and in the third month after injection. The study was planned as a randomized controlled prospective study.

DETAILED DESCRIPTION:
Patients diagnosed with epicondylitis in our outpatient clinic will be divided into 3 groups, and patients who will receive saline in 1 group and betamethasone sodium in a group will be selected in accordance with the specified conditions and their treatment will be started, and the treatment will be started, which patient will receive which treatment will be determined by the computerized randomization program. ), 1ml prp (plate-rich plasma to be prepared with the blood taken from the patient on the day of injection), 1 ml saline (0.9 NACI), while the patient is in the supine position, the affected elbow is 90 flexion and neutral rotation, The non-dominant thumb will be placed at the sensitive point in the lateral epicondyle. The injection will be applied to the point with a 23 g needle. After the injection, the subjects will be taught a stretching exercise of the joint extensors of the wrist and fingers. Subjects will be asked to do this exercise five times in one session, two sessions a day.Examination and functional scores to be applied to the patients during follow-up: VAS, DASH and PRTEE scores will be checked in the 1st 6th week, 3rd month, 6th month and 12th month VAS: Visual Analog Scale DASH: The Disabilities of the Arm, Shoulder and Hand PRTEE: The Patient-Rated Tennis Elbow Evaluation 2. It will be evaluated by USG in the 3rd month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18
2. Clinical diagnosis-
3. Symptoms lasting more than 3 months and no injection within this period
4. Radiologically diagnosed -

Exclusion Criteria:

- 1. symptoms for less than 3 months 2. Having been given injection treatment within 3 months

3. Surgical procedure for lateral epicondylitis 4. Having pain caused by the cervical spine 5. Restricted elbow range of motion 6.Having an elbow bony deformity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
CHANGE İN VAS: Visual Analog Skala | baseline and 6th week, 3rd month, 6th month and 12th month
  we ask questions for vas score ıt has explained https://www.orthopaedicscore.com/, minum score 1 maximum 10 The higher the score, the greater the pain, and we expect it to decrease after the process.
CHANGE İN DASH: The Disabilities of the Arm, Shoulder and Hand | baseline and 6th week, 3rd month, 6th month and 12th month
  we ask questions which has explained in https://www.orthopaedicscore.com/ The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability)-this is called the DASH score. we expect it to decrease after the process.
CHANGE İN PRTEE: The Patient-Rated Tennis Elbow Evaluation | baseline and 6th week, 3rd month, 6th month and 12th month
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is designed to evaluate pain and disability in subjects with lateral elbow tendinopathy. This questionnaire is available in Swedish, Italian, and some other languages. A Persian language version of the questionnaire is needed for both research and clinical purposes. The higher the score, the greater the pain, and we expect it to decrease after the process.

SECONDARY OUTCOMES:
evaluation common extensor morphology and vascularity with ultrasound | baseline and 3 months after enjection
  ıt will perform by radiology doctor in istanbul university radiology department , In order to assess common extensor tendon morphology and vascularity, ana-tomic grayscale US images of the injected elbow wereperformed to establish the degree of tendinosis, using anL17-5 linear-phased transducer (Philips Medical Systems,Bothell, WA, USA) with the elbow in flexion and forearmpronated to the "thumbs up"position. Contrast harmonicimaging, using an amplitude modulation technique, wasperformed with the patient sitting and the elbow in flexionusing an L12-5 phased-array linear transducer with an IU22US scanner (Phillips Medical Systems, Bothell, WA, USA)to visualize the common extensor tendon at the lateralepicondyle

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaudhury S, de La Lama M, Adler RS, Gulotta LV, Skonieczki B, Chang A, Moley P, Cordasco F, Hannafin J, Fealy S. Platelet-rich plasma for the treatment of lateral epicondylitis: sonographic assessment of tendon morphology and vascularity (pilot study). Skeletal Radiol. 2013 Jan;42(1):91-7. doi: 10.1007/s00256-012-1518-y. Epub 2012 Sep 22. PMID 23001116
- [Result] Wolf JM, Ozer K, Scott F, Gordon MJ, Williams AE. Comparison of autologous blood, corticosteroid, and saline injection in the treatment of lateral epicondylitis: a prospective, randomized, controlled multicenter study. J Hand Surg Am. 2011 Aug;36(8):1269-72. doi: 10.1016/j.jhsa.2011.05.014. Epub 2011 Jun 25. PMID 21705157
- See also: https://www.sciencedirect.com/science/article/abs/pii/S0363502311006289 — https://pubmed.ncbi.nlm.nih.gov/21705157/